CLINICAL TRIAL: NCT02270164
Title: The Impact of Artichoke Leaf Extract on Blood Cholesterol: Primary Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor discontinued funding due to higher than anticipated manufacturer costs
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Indena S.p.A (Industry)
Responsible Party: Principal Investigator, Daniel Riche, Associate Professor, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2014-0167
Record Dates: First submitted 2014-10-09; First posted 2014-10-21 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Lipid Metabolism Disorders
Keywords: Lipids; Cholesterol; Dietary Supplements; Cynara scolymus; Safety
MeSH Terms: conditions — Lipid Metabolism Disorders | interventions — artichoke leaf

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Artichoke Leaf Extract (Experimental): Pycrinil® 100 mg/flaxseed oil 380 mg liquid filled hard plant based capsules (Licaps®) twice daily with food
  Interventions: Dietary Supplement: Artichoke Leaf Extract
- Placebo (Placebo Comparator): Placebo/flaxseed oil 380 mg liquid filled hard plant based capsules (Licaps®) twice daily with food
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Artichoke Leaf Extract — Capsule
  Other Names: Pycrinil
  Arms: Artichoke Leaf Extract
Other: Placebo — Capsule
  Arms: Placebo

SUMMARY:
Pycrinil® is a purified extract of the artichoke leaf. Artichoke leaf extract (ALE) has some clinical trial data suggesting benefit in the treatment of cholesterol disorders in several countries, but this effect has not been studied in a U.S. population. The investigators will give ALE or a placebo to overweight men and women with low "good" cholesterol to see if ALE increases their good cholesterol. The investigators will also make sure that ALE is safe.

DETAILED DESCRIPTION:
Subjects will be divided into one of two groups: (1) Pycrinil®/flaxseed oil or (2) Placebo/flaxseed oil twice daily with food. The two formulations will be identical in appearance and standardized by Indena, S.p.A. Patients will be enrolled for a total of 3 months (± 1 week to allow for scheduling flexibility) with a 1 month (± 1 week to allow for scheduling flexibility) first follow-up visit in between enrollment and final visits. At all visits, patients will be asked to monitor for any symptomatic ADE. The first follow-up visit will focus on medication compliance (via pill count) and safety assessment (including laboratories). The final study visit will consist of brief clinical assessment (including anthropometrics), completed lifestyle and physical activity assessments, subjective ADE reporting, and donated blood and urine for clinical laboratory tests. Medication changes are not prohibited during the study period, but must be recorded. Medication bottles will be collected at the first follow-up and final visits; pill counts will be performed to assess compliance.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* HDL cholesterol <40 mg/dL in men or <50 mg/dL in women
* BMI ≥25 kg/m2.

Exclusion Criteria:

* Patient on statins
* Triglycerides >400 mg/dL
* Low density lipoprotein (LDL) >190 mg/dL
* Significant hepatic disease (i.e., documented diagnosis of hepatic cancer, hepatitis, or cirrhosis)
* Significant renal disease (i.e., most recent glomerular filtration rate <30 mL/min/1.73 m2)
* Significant gastrointestinal tract disease (documented diagnosis of malabsorption disorder, GI cancer, or uncontrolled inflammatory bowel disease)
* History of transplant
* Women of reproductive potential not receiving birth control
* Pregnant/nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in Concentrations of High Density Lipoprotein Cholesterol | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Riche, PharmD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

REFERENCES:
- [Background] Bundy R, Walker AF, Middleton RW, Wallis C, Simpson HC. Artichoke leaf extract (Cynara scolymus) reduces plasma cholesterol in otherwise healthy hypercholesterolemic adults: a randomized, double blind placebo controlled trial. Phytomedicine. 2008 Sep;15(9):668-75. doi: 10.1016/j.phymed.2008.03.001. PMID 18424099
- [Background] Englisch W, Beckers C, Unkauf M, Ruepp M, Zinserling V. Efficacy of Artichoke dry extract in patients with hyperlipoproteinemia. Arzneimittelforschung. 2000 Mar;50(3):260-5. doi: 10.1055/s-0031-1300196. PMID 10758778
- [Background] Rondanelli M, Giacosa A, Opizzi A, Faliva MA, Sala P, Perna S, Riva A, Morazzoni P, Bombardelli E. Beneficial effects of artichoke leaf extract supplementation on increasing HDL-cholesterol in subjects with primary mild hypercholesterolaemia: a double-blind, randomized, placebo-controlled trial. Int J Food Sci Nutr. 2013 Feb;64(1):7-15. doi: 10.3109/09637486.2012.700920. Epub 2012 Jun 29. PMID 22746542
- [Background] Wider B, Pittler MH, Thompson-Coon J, Ernst E. Artichoke leaf extract for treating hypercholesterolaemia. Cochrane Database Syst Rev. 2013 Mar 28;(3):CD003335. doi: 10.1002/14651858.CD003335.pub3. PMID 23543518